CLINICAL TRIAL: NCT05025280
Title: Sensory Processing Patterns in Adults With Acquired Hearing Loss
Brief Title: Sensory Processing Patterns in Hearing Loss
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Bilgehan Tekin Dal, Principal Investigator, Gazi University
Other Study IDs: 5057087197
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hearing Loss
Keywords: Adult; Hearing loss; sensory processing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hearing loss: According to the audiological test results, individuals with a pure tone average of more than 25 dB in the better ear and with less than 10 dB difference between the air-bone conduction thresholds
  Interventions: Other: Adolescent/Adult Sensory Profile Questionnaire
- normal hearing: According to the audiological test results, individuals with a pure tone average of 25 dB or less in both ears and with less than 10 dB difference between the air-bone conduction thresholds
  Interventions: Other: Adolescent/Adult Sensory Profile Questionnaire

INTERVENTIONS:
Other: Adolescent/Adult Sensory Profile Questionnaire — The Adolescent/Adult Sensory Profile Questionnaire (AASP), was developed based on Dunn's model of sensory processing. It is a 60-item self-assessment questionnaire that evaluates behavioral patterns related to sensory processing. The questionnaire consists of six different subsections such as taste/smell processing, movement processing, visual processing, touch processing, auditory processing, and activity level. According to the answers given, individuals are evaluated in 4 quartiles as "low registration," "sensory sensitivity," "sensation avoiding," and "sensation seeking."

SUMMARY:
This study aimed to evaluate the sensory processing abilities of adults with acquired hearing loss and to explore the differences in sensory processing between adults with hearing loss and adults with normal hearing. Sensory processing functions of 30 adults with acquired hearing loss will be evaluated using the Adolescent/Adult Sensory Profile. The data from adults with hearing loss will be compared with data from 30 adults with normal hearing who were similar in gender and age.

DETAILED DESCRIPTION:
This study aims to investigate the sensory processing patterns of adults with hearing loss and compare them with healthy controls. In this study, it was hypothesized that adults with hearing loss, had an abnormal sensory profile like children with hearing loss.

Participants will consist of individuals between the ages of 18-65 who were taken into audiological evaluation at the outpatient unit of Audiology of a hospital and voluntarily agreed to participate in the study.

According to the audiological test results, individuals with a pure tone average of more than 25 decibel (dB) in the better ear and with less than 10 dB difference between the air-bone conduction thresholds will be included in the study group, and those with a pure tone average of 25 dB or less in both ears and with less than 10 dB difference between the air-bone conduction thresholds will be included in the control group.

Hearing aid users, those with chronic tinnitus and/or dizziness, and those with major medical disorders and/or handicaps will not be included in the study. In this study, Hearing Handicap Inventory for Adults (HHIA) and Adolescent/Adult Sensory Profile will be used.

ELIGIBILITY:
Inclusion Criteria:

* adults with acquired sensorineural hearing loss for study group
* adults with normal hearing for control group

Exclusion Criteria:

* Hearing aid users
* adults with chronic tinnitus and/or dizziness
* adults with major medical disorders and/or handicap

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the audiological test results, individuals with a pure tone average of more than 25 dB in the better ear and with less than 10 dB difference between the air-bone conduction thresholds
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Adolescent/Adult Sensory Profile scores | 6 months
  There are 15 questions in each quadrant for 60 questions in total. The responses provided are in a Likert-scale system with "almost always (5 points)", "often", "sometimes", "rarely" and "almost never (1 point)" and the scores of the related items are summed up to provide the score for each quadrant. Norm values have been established for three different age intervals: 11-18, 18-65, and 65 years and over for evaluation and respondents are classified in the end for the four quadrants using the statements "much more than most people," "more than most people," "similar to most people," "less than most people," and "much less than most people".
  Respectively Sensory Processing Reference Ranges (18-64 yr)
  * Low registration 15-18, 19-23, 24-35, 36-44, 45-75
  * Sensation seeking 15-35, 36-42, 43-56, 57-62, 63-75
  * Sensory sensitivity 15-18, 19-25, 26-41, 42-48, 49-75
  * Sensation avoiding 15-19, 20-26, 27-41, 42-49, 50-75

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participant data are not to be shared with other researches